CLINICAL TRIAL: NCT02594397
Title: Acupuncture for Diabetic Gastroparalysis: a Randomized Controlled Trial
Acronym: ADG-RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Hunan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014CB543102-2
Record Dates: First submitted 2015-10-31; First posted 2015-11-03 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-09

CONDITIONS: Gastroparesis; Diabetes Complications
MeSH Terms: conditions — Gastroparesis; Diabetes Complications

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (3):
- acupoints combination 1 (Experimental): acupoints comination 1 includes the specific acupoint ST36 (Zusanli) and a local acupoint CV12 (Zhongwan).
  Interventions: Other: acupoints combination 1
- acupoints combination 2 (Active Comparator): acupoints comination 2 includes the specific acupoint ST36 (Zusanli) and a distal acupoint PC6(Neiguan).
  Interventions: Other: acupoints combination 2
- sham acupoints combination (Sham Comparator): sham acupoints combination includes the specific acupoint ST36 (Zusanli) and a sham acupoint.
  Interventions: Other: sham acupoints combination

INTERVENTIONS:
Other: acupoints combination 1
  Arms: acupoints combination 1
Other: acupoints combination 2
  Arms: acupoints combination 2
Other: sham acupoints combination
  Arms: sham acupoints combination

SUMMARY:
The purpose of this study is to determine whether the different combination of acupoints have different effect on diabetic gastroparalysis.

ELIGIBILITY:
Inclusion Criteria:

* individuals who meet the diagnostic criteria of diabetes gastric paralysis.
* individuals between the ages of 18 and 60 years.
* individuals who meet blood glucose control standards: Fasting plasma glucose (FPG) ≤7. 8mmol/L; 2 hours plasma glucose (2hPG)≤13.6mmol/L.
* individuals who suffered for more than 3 years.
* individuals who treated with diet control or exercise or using hypoglycemic drug (except for α-glucosidase Inhibitor) on the basis of diet or exercise therapy and the dose stability must be last at least 3 months.
* individuals who receive no other treatments in the first 3 months.
* women who is at the age of childbearing age and take contraceptive measures.
* individuals who voluntarily agree with a study protocol and sign a written informed consent.

Exclusion Criteria:

* individuals who have reflux esophagitis;
* individuals who have gastroparesis after surgery;
* individuals who have acute complications with ketoacidosis and nonketotic hyperosmolar coma;
* individuals who have Acute cardiovascular and cerebrovascular diseases or Severe trauma or surgery, severe infection. Or who are pregnant or breastfeeding;
* individuals who have a history disease of myocardial infarction, acute coronary syndrome or coronary revascularization;
* individuals who have serious hepatobiliary disease, or AST and/or ALT 2 times greater than the upper limit of normal patients;
* individuals with kidney damage, and serum creatinine exceeds 140umol/L;
* individuals who have obvious blood system diseases (Any one of which can not be caught in line: Hb: male<110g/L, women<100g/L,WBC<3.5×109/L,PLT<80×109/L).
* individuals who have a problem of blood press:SBP≥180mmHg,DPB≥100mmHg;
* individuals who have cancer or other serious progressive wasting disease, and easy to infection and bleeding;
* individuals who have peptic ulcer or other organic disease confirmed by esophagogastroduodenoscopy;
* individuals unwilling to meet the testing and exacerbations,or have serious complications in the test;
* individuals who have taking α-glucosidase inhibitor drug in the past four weeks.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
the score of GCSI | 4 weeks
  GCSI means gastroparesis cardinal symptom index

SECONDARY OUTCOMES:
Gastric emptying time | 4 weeks
gastrin concentrations | 4 weeks
motilin concentrations | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zenghui Yue, Prof., Study Chair — Hunan University of Chinese Medicine

REFERENCES:
- [Derived] Xuefen W, Ping L, Li L, Xiaoli C, Yue Z. A Clinical Randomized Controlled Trial of Acupuncture Treatment of Gastroparesis Using Different Acupoints. Pain Res Manag. 2020 Apr 25;2020:8751958. doi: 10.1155/2020/8751958. eCollection 2020. PMID 32399130